CLINICAL TRIAL: NCT07356388
Title: An Study on the Efficacy and Safety of Finerenone in Proteinuria Patients After Kidney Transplantation
Brief Title: FINEPKT - Finerenone in Proteinuria Patients After Kidney Transplan
Acronym: FINEPKT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: kewen Chen,MD (Other)
Responsible Party: Sponsor-Investigator, kewen Chen,MD, Attending Physician, First Affiliated Hospital of the Chinese People's Liberation Army Naval Medical University
Organization: First Affiliated Hospital of the Chinese People's Liberation Army Naval Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHEC2024-255
Record Dates: First submitted 2025-12-17; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Kidney Transplantation Recipients; Proteinuria Patients
Keywords: proteinuria patients; kidney transplantation; Finerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Experimental Group — Oral ACEI/ARB (e.g., valsartan capsules 80mg qd or 150mg qd) + finelidone (10 or 20mg orally once a day)
Drug: Control (Standard treatment) — Oral ACEI/ARB (e.g., valsartan capsules 80mg qd or 150mg qd) + Dapagliflozin (10 or 20mg orally once a day)

SUMMARY:
The goal of this clinical trial is to learn if Finerenone works to treat proteinuria patients after kidney transplantation. It will also learn about the safety of Finerenone. The main questions it aims to answer are:

Does Finerenone lower the number of UACR values in kidney transplant recipients?? What medical problems do participants have when taking Finerenone? Researchers will compare Finerenone to Dapagliflozin to see if Finerenone works to treat proteinuria patients after kidney transplantation.

DETAILED DESCRIPTION:
This project is designed as a single-center, prospective, randomized controlled clinical study with strict inclusion and exclusion criteria. Based on statistical sample size estimation, it aims to enroll kidney transplant recipients with proteinuria, collect basic clinical data of the recipients, and monitor primary and secondary efficacy indicators after transplantation, with the establishment of warning events. The study will further evaluate the long-term clinical benefits of Finerenone in patients with proteinuria after kidney transplantation, in order to formulate better medication plans and provide an ideal reference for similar cases (such as elevated blood creatinine after kidney transplantation).

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult kidney transplant patients (≥18 years old) 2. The diagnosis and screening of chronic kidney disease (CKD) after kidney transplantation meet at least one of the following criteria:

  1. Persistent high proteinuria (UACR of 30-300 mg/g, more than 2 of 3 early morning urination samples) and estimated glomerular filtration rate (eGFR) of 25-60ml/min/1.73m2 (CKD EPI) and the presence of diabetic retinopathy.
  2. Persistent extremely high albuminuria (UACR≥300mg/g, more than 2 of 3 early morning urination samples) and eGFR≤25 mL /min/1.73m2 (CKD EPI) 3. Previous treatments with angiotensin-converting enzyme inhibitors (ACEI) and angiotensin receptor block (ARB) are as follows: A. At least 4 weeks prior to the run-in visit, subjects should receive ACEI or ARB or a combination of both

  b. At the beginning of the run-in visit, subjects were receiving only ACEI or ARB or a combination of both.

  c. At least 4 weeks prior to the screening visit, subjects should be treated with only the maximum tolerated labeled dose (but not less than the minimum labeled dose) of ACEI or ARB, preferably without adjustment of dose or drug selectivity or any other antihypertensive or antiglycemic therapy.

  4. Serum potassium ≤4.8mmol/L during running-in and screening. 5. Voluntarily sign informed consent

Exclusion Criteria:

* 1. Kidney transplant recipients have a history of retransplantation, multiple kidney transplants, and transplantation of other organs and tissues.

  2. Known significant non-diabetic nephropathy, including clinically relevant renal artery stenosis.

  3. Uncontrolled arterial hypertension (i.e. mean sitting systolic blood pressure (SBP) ≥170mmHg at presentation, sitting diastolic blood pressure (DBP) ≥110mmHg, or mean sitting SBP≥160mmHg, sitting DBP≥ 100mmHg at screening) 4. In patients with type I diabetes, the hemoglobin a1C (HbA1c) is >12%. 5. Uncontrolled hypotension; The mean SBP at run-in visit or screening visit was <90mmHg 6. Chronic heart failure clinically diagnosed at run-in visit with decreased ejection fraction (HFrEF) and persistent symptoms (New York Heart Association [NYHA] Grade II-IV) (Level 1A recommendation for salocorticoid receptor antagonist MRA) 7. Hospitalization for stroke, transient ischemic attack, acute coronary syndrome, or worsening heart failure within 30 days prior to screening 8. Hemokalium was higher than 5.5mmol/L within 12 weeks after treatment due to acute renal failure 9. Patients with malignant tumors or other metabolic disorders have a history of allergic diseases or allergies 10. Severe liver damage 11 Pregnant or lactating women 12. Severe infectious diseases 13. There are other circumstances that the investigator deems inappropriate to participate in the clinical trial.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Urine Albumin-to-Creatinine Ratio | From enrollment to the end of treatment at 6 months"
creatinine | From enrollment to the end of treatment at 6 months"

SECONDARY OUTCOMES:
24h UTP | From enrollment to the end of treatment at 6 months"
  24-hour Urinary Total Protein
eGFR | From enrollment to the end of treatment at 6 months"

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barrera-Chimal J, Lima-Posada I, Bakris GL, Jaisser F. Mineralocorticoid receptor antagonists in diabetic kidney disease - mechanistic and therapeutic effects. Nat Rev Nephrol. 2022 Jan;18(1):56-70. doi: 10.1038/s41581-021-00490-8. Epub 2021 Oct 21. PMID 34675379
- [Background] Al Dhaybi O, Bakris GL. Non-steroidal mineralocorticoid antagonists: Prospects for renoprotection in diabetic kidney disease. Diabetes Obes Metab. 2020 Apr;22 Suppl 1:69-76. doi: 10.1111/dom.13983. PMID 32267074
- [Background] Kolkhof P, Joseph A, Kintscher U. Nonsteroidal mineralocorticoid receptor antagonism for cardiovascular and renal disorders - New perspectives for combination therapy. Pharmacol Res. 2021 Oct;172:105859. doi: 10.1016/j.phrs.2021.105859. Epub 2021 Aug 28. PMID 34461222
- [Background] Filippatos G, Bakris GL, Pitt B, Agarwal R, Rossing P, Ruilope LM, Butler J, Lam CSP, Kolkhof P, Roberts L, Tasto C, Joseph A, Anker SD; FIDELIO-DKD Investigators. Finerenone Reduces New-Onset Atrial Fibrillation in Patients With Chronic Kidney Disease and Type 2 Diabetes. J Am Coll Cardiol. 2021 Jul 13;78(2):142-152. doi: 10.1016/j.jacc.2021.04.079. Epub 2021 May 17. PMID 34015478
- [Background] Bakris GL, Agarwal R, Chan JC, Cooper ME, Gansevoort RT, Haller H, Remuzzi G, Rossing P, Schmieder RE, Nowack C, Kolkhof P, Joseph A, Pieper A, Kimmeskamp-Kirschbaum N, Ruilope LM; Mineralocorticoid Receptor Antagonist Tolerability Study-Diabetic Nephropathy (ARTS-DN) Study Group. Effect of Finerenone on Albuminuria in Patients With Diabetic Nephropathy: A Randomized Clinical Trial. JAMA. 2015 Sep 1;314(9):884-94. doi: 10.1001/jama.2015.10081. PMID 26325557
- [Background] Filippatos G, Anker SD, Agarwal R, Pitt B, Ruilope LM, Rossing P, Kolkhof P, Schloemer P, Tornus I, Joseph A, Bakris GL; FIDELIO-DKD Investigators. Finerenone and Cardiovascular Outcomes in Patients With Chronic Kidney Disease and Type 2 Diabetes. Circulation. 2021 Feb 9;143(6):540-552. doi: 10.1161/CIRCULATIONAHA.120.051898. Epub 2020 Nov 16. PMID 33198491
- [Background] Pitt B, Filippatos G, Agarwal R, Anker SD, Bakris GL, Rossing P, Joseph A, Kolkhof P, Nowack C, Schloemer P, Ruilope LM; FIGARO-DKD Investigators. Cardiovascular Events with Finerenone in Kidney Disease and Type 2 Diabetes. N Engl J Med. 2021 Dec 9;385(24):2252-2263. doi: 10.1056/NEJMoa2110956. Epub 2021 Aug 28. PMID 34449181
- [Background] Bakris GL, Agarwal R, Anker SD, Pitt B, Ruilope LM, Rossing P, Kolkhof P, Nowack C, Schloemer P, Joseph A, Filippatos G; FIDELIO-DKD Investigators. Effect of Finerenone on Chronic Kidney Disease Outcomes in Type 2 Diabetes. N Engl J Med. 2020 Dec 3;383(23):2219-2229. doi: 10.1056/NEJMoa2025845. Epub 2020 Oct 23. PMID 33264825